CLINICAL TRIAL: NCT06809985
Title: Latent Phase Membrane Stripping for Caesarean Section Reduction. Single Blind Clinical Trial
Brief Title: Latent Phase Membrane Stripping for Caesarean Section Reduction
Acronym: DEMEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PGO-UNAH-48-6-2025
Record Dates: First submitted 2025-01-15; First posted 2025-02-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Delivery; Cervical Ripening; Latent Phase Labour
Keywords: Cesarean Delivery; Cervical ripening; latent phase labour; hamilton maneuver

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, efficacy, superiority, single-blind clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Both the patient and the principal investigator will know the intervention, the data analyst researcher does not know the group to which the patients have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hamilton maneuver (Experimental): The Hamilton maneuver is performed by inserting one or two fingers through the internal cervical os and carefully producing a circumferential rotational movement through the uterine segment in order to separate the fetal membranes from the decidua. This maneuver is recommended in order to reduce the need for formal induction.
  Interventions: Procedure: Hamilton maneuver
- Control (No Intervention): A normal gynecological evaluation will be performed, no additional maneuvers will be performed in addition to the routine evaluation of the patient.

INTERVENTIONS:
Procedure: Hamilton maneuver — The Hamilton maneuver is performed by inserting one or two fingers through the internal cervical os and carefully producing a circumferential rotational movement through the uterine segment in order to separate the fetal membranes from the decidua. This maneuver is recommended in order to reduce the need for formal induction.
  Other Names: membrane decollege; membrane sweep
  Arms: Hamilton maneuver

SUMMARY:
In the Hospital Escuela, the availability of beds and criteria for admission to the intensive care unit ICU are not the same, the use of this marker is questionable, as it is affected by the level of complexity of care provided to a health setting and the organization of obstetric care. The cesarean section rate (almost 63.2%), is without significant variation by different criteria.

The importance of finding strategies to reduce the rate of cesarean births and thus counteract the high rates of maternal morbidity and mortality is proposed. For this reason, this research is aimed at reducing the latent phase of labor through the use of the Hamilton maneuver.

DETAILED DESCRIPTION:
There is a need to find non-pharmacological interventions that can speed up delivery to prevent maternal complications and reduce the number of caesarean sections.

Maternal mortality remains one of the biggest health problems worldwide. Every day, around 830 women die worldwide from complications related to pregnancy or childbirth. In 2015, an estimated 303,000 women died during pregnancy and childbirth or after. Most of these deaths occur in low-income countries and most of them could have been prevented. The maternal mortality rate in Latin American and Caribbean countries, calculated by the Inter-Agency Group (MMEIG), shows a significant decrease as a regional average in recent years, from 88 per 100,000 live births in 2005 to 67 per 100,000 live births in 2015.

At the Escuela Hospital, the availability of beds and admission criteria in the intensive care unit (ICU) are not the same. The use of this marker is questionable, since it is affected by the level of complexity of the care provided to a health setting and the organization of obstetric care. We found in our study a cesarean section rate (almost 63.2%), with no significant variation by different criteria. This finding is consistent with that reported by Nelissen et al. Due to the severity of the obstetric conditions of these patients, their pregnancy usually requires urgent action. Although cesarean section is associated with high rates of maternal morbidity and mortality compared to vaginal delivery, when clinically indicated, timely termination of pregnancy can reduce the risk of maternal-fetal death.

Based on the above, this research proposes the importance of finding strategies to reduce the rate of cesarean deliveries and thus counteract the high rates of maternal morbidity and mortality. For this reason, this research is aimed at reducing the latent phase of labor through the use of the Hamilton maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Submission of a signed and dated informed consent form.
* Declared willingness to comply with all study procedures and availability for the duration of the study.
* nulliparous
* woman with singleton pregnancy at 37 weeks or more
* integral membranes
* cephalic presentation
* Bishop's score less than 7
* No contraindication for vaginal delivery

Exclusion Criteria:

* Previous uterine surgery
* Maternal condition preventing vaginal delivery
* Fetal anomaly
* Premature rupture of membranes
* Multiple pregnancy
* Fetal orbit
* Myomas
* Maternal comorbidities such as chronic arterial hypertension, type 1, 2 and gestational diabetes, hypothyroidism, among others.
* Anemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Time from admission until active phase | Since intervention until 20 hours
  time from the intervention to reach a cervical dilatation greater than or equal to 5 cm

SECONDARY OUTCOMES:
Rate of cesarean births | Since intervention until 7 days or maternal discharge
  number of cesarean sections in the patients
Level of Maternal satisfaction | Since intervention until 24 hours of delivery or maternal discharge
  For the evaluation of the perception of support and birth control, the Mackey MSCRS scale will be used, with a baseline assessment when the patient has cervical dilatation between 0 and 3 cm and a second assessment 24 hours after delivery, there are 35 items, likert scale type, For the evaluation of the perception of support and birth control, the Mackey MSCRS scale will be used, with a baseline assessment when the patient has cervical dilatation between 0 and 3 cm and a second assessment 24 hours after delivery.
Rate of maternal complications | Since intervention until 14 days
  Signs of maternal complications as fever, endometritis

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc., Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Finucane EM, Murphy DJ, Biesty LM, Gyte GM, Cotter AM, Ryan EM, Boulvain M, Devane D. Membrane sweeping for induction of labour. Cochrane Database Syst Rev. 2020 Feb 27;2(2):CD000451. doi: 10.1002/14651858.CD000451.pub3. PMID 32103497